CLINICAL TRIAL: NCT03977922
Title: A Pilot Nutrition Program for Spinal Cord Injury and MS: Effects on Inflammation, Cardiometabolic Health and Psychosocial Well-being
Brief Title: A Pilot Nutrition Program for Spinal Cord Injury and MS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brock University (Other)
Responsible Party: Principal Investigator, David Ditor, Professor, Kinesiology, Brock University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18-309 - Ditor
Record Dates: First submitted 2019-06-05; First posted 2019-06-06 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Spinal Cord Injuries; Multiple Sclerosis
MeSH Terms: conditions — Spinal Cord Injuries; Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diet group (Experimental): The diet group will be involved in a 12-week pilot nutrition program based on the anti-inflammatory diet studied by Allison and Ditor (2015). The nutrition program will entail:
  1. Once per week (Monday mornings), nutrition program members will come to Power Cord to pick up their box of ingredients for their meals that week (Monday to Friday). Recipe cards will accompany the ingredients, and enough food will be provided for 3 meals and 2 snacks per day. The meals will be based on the anti-inflammatory diet previously studied in Allison and Ditor (2015).
  2. 10-12 online videos that cover basic kitchen/cooking skills, how to prepare the meals in the program, how to shop for healthy foods at the grocery store, etc.
  3. At the beginning of the program each member will be provided with a few pieces of accessible kitchen equipment that will made food preparation and cooking much easier.
  4. Once per month, we will be offering a live cooking class.
  Interventions: Other: Diet group
- Control group (No Intervention): The control group will eat their usual diet for the 12-week period.

INTERVENTIONS:
Other: Diet group — The diet group will be involved in a 12-week pilot nutrition program that will be based on the anti-inflammatory diet previously studied by Allison and Ditor (2015).
  Arms: Diet group

SUMMARY:
The purpose of this study is to determine the feasibility of a 12-week pilot community-based nutrition program for individuals with spinal cord injury and multiple sclerosis, and to determine the effects of the nutrition program on body composition, inflammation, neuropathic pain, depression and quality of life.

DETAILED DESCRIPTION:
Spinal cord injury (SCI) and multiple sclerosis (MS) are both conditions characterized by chronic inflammation as indicated by elevated levels of circulating pro-inflammatory cytokines. These cytokines can have a wide array of negative impacts in the body. For example, pro-inflammatory cytokines can impair serotonin production and usage in the brain and thus increase the risk of depression. Likewise, they can sensitize nociceptors and increase the intensity and frequency of neuropathic pain. Recent work has shown that a 3-month anti-inflammatory diet is not only effective in reducing pro-inflammatory cytokines, but also reduced self-reported depression and neuropathic pain, by approximately 55% and 40%, respectively (Allison and Ditor, 2015; Allison et al., 2016). These data are very promising since both depression and neuropathic pain are highly prevalent after SCI and MS, and current pharmacological treatments are only partially effective and associated with unwanted side-effects.

Despite the highly encouraging results mentioned above, one year following the conclusion of the study participants were no longer adhering to the anti-inflammatory diet. Specifically, during the actual study, adherence to the diet was, on average 89% (70-100%), while at one-year follow-up, adherence fell to, on average 43% (36-53%), which was virtually the same as baseline eating habits (Allison and Ditor, 2018). Likewise, measures of depression went back to baseline as well. These follow-up data prompted a subsequent qualitative study in which former participants were interviewed as a means to identify the facilitators and barriers that affect one's ability to adhere to the anti-inflammatory diet (Bailey et al., 2018). This qualitative study is now being used to inform a nutrition program that is in the early stages of development at a wheelchair accessible exercise facility; Power Cord.

The nutrition program will consist of 4 aspects:

1. Once per week (Monday mornings), nutrition program members will come to Power Cord to pick up their box of ingredients for their meals that week (Monday to Friday). Recipe cards will accompany the ingredients, and enough food will be provided for 3 meals and 2 snacks per day. The meals will be based on the anti-inflammatory diet mentioned above. The nutrition program will not provide ingredients for Saturdays and Sundays, for three reasons. First, research has shown that occasional "cheat meals" help with long term compliance to the diet. Second, members should eventually become self-sufficient and even wean themselves off the nutrition program (or reduce their involvement). Third, this reduces the cost of the program and will help with long term sustainability.
2. To assist the members with meal preparation, there will also be 10-12 online videos that cover basic kitchen/cooking skills, how to prepare the meals in the program, how to shop for healthy foods at the grocery store, etc.
3. At the beginning of the program each member will be provided with a few pieces of accessible kitchen equipment that will made food preparation and cooking much easier. The equipment includes, a 1 Second Slicer (to be used in place of a knife), a padded lap tray (to be used as a cutting surface on the lap instead of a counter), a toaster oven, light weight pots and pans, a Nutri Bullet Blender.
4. Once per month, there will be a live cooking class.

Before this nutrition program can be long-term and sustainable, a 12-week pilot program will be completed to help determine the eventual membership pricing and feasibility. This pilot will also be used to determine the effects of the diet on body composition, inflammation, neuropathic pain, depression and quality of life. This pilot program will include 15 existing Power Cord members; 5 with SCI and 5 with MS who will be in the diet group, and 5 individuals with SCI and MS who will serve as controls. Participants in the pilot program will only pay $100/month for their involvement, and this will include their kitchen equipment, food for the 3-months, cooking classes and access to online content. The study and outcome measures described in this posting pertain to the 3-month pilot nutrition program.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with spinal cord injury may be of any level of injury (paraplegia/tetraplegia) and severity of injury (complete/incomplete) and will be at least one year post-injury.
* Individuals with MS will have a diagnosis of relapsing remitting MS or secondary progressive MS, and will be at least one year post-diagnosis.

Exclusion Criteria:

* . Participants will be asymptomatic for pressure ulcers, urinary tract infections or respiratory infections at the time of recruitment, and they may be recreationally active but those participating in elite or high-level athletics/training will be excluded from the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2022-02-28 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Change from baseline body composition at 12 weeks | Before and after the 12-week nutrition program (in both groups)
  Dual-energy x-ray absorptiometry (DEXA) to measure the percentage of body fat.
Change from baseline inflammation at 12 weeks | Before and after the 12-week nutrition program (in both groups)
  Blood samples will be analyzed for various inflammatory mediators
Change from baseline neuropathic pain at 12 weeks | Before and after the 12-week nutrition program (in both groups)
  The Neuropathic pain questionnaire will be used to determine self-reported neuropathic pain
Change from baseline depression at 12 weeks | Before and after the 12-week nutrition program (in both groups)
  The Center for Epidemiological Studies Depression scale (CES-D) will be used to determine self-reported depression. This scale ranges from 0 to 60 with higher scored indicating more depression.
Change from baseline perceived quality of Life at 12 weeks | Before and after the 12-week nutrition program (in both groups)
  The Perceived Quality of Life questionnaire (PQOL) will be used to determine self-reported quality of life
Change from baseline blood lipids at 12 weeks | Before and after the 12-week nutrition program (in both groups)
  Blood samples will be analyzed for blood lipids
Change from baseline glucose tolerance at 12 weeks | Before and after the 12-week nutrition program (in both groups)
  Blood samples will be analyzed for HbA1c

SECONDARY OUTCOMES:
Dietary intake | At baseline, and after 4 weeks, 8 weeks and 12 weeks (in both groups)
  Food logs will be collected to determine adherence to the dietary intake during the 12-week study for both groups.

CONTACTS AND LOCATIONS:
Overall Officials: David S Ditor, PhD, Principal Investigator — Brock University
Locations (1):
- Brock University, Saint Catharines, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No